CLINICAL TRIAL: NCT03908983
Title: OPtimisation of Surgical Repair for Treating Insufficiency of the MItral Valve - Safety and Effectiveness Evaluation (OPTIMISE II)
Brief Title: OPtimisation of Surgical Repair for Treating Insufficiency of the MItral Valve - Safety and Effectiveness Evaluation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kephalios (Industry)
Responsible Party: Sponsor
Organization: Affluent Medical (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPTIMISE II
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Mitral Valve Regurgitation
Keywords: Mitral Regurgitation; Mitral valve repair; Mitral annuloplasty; Adjustable annuloplasty
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implanted Patients (Experimental): Implantation of Kalios Device
  Interventions: Device: Kalios Implant

INTERVENTIONS:
Device: Kalios Implant — KALIOS is an adjustable annuloplasty ring, to be implanted by open surgery, having a hollow structure that comprises a flat rigid ring surrounding a deformable cage. The unique feature of KALIOS is that its annular shape and dimension can be finely adjusted percutaneously by an external actuator (three-balloon catheter) independently in the three areas corresponding to P1, P2 and P3

SUMMARY:
KALIOS is indicated for the surgical treatment of mitral regurgitation by mitral valve repair.It is intended for mitral valve repair using conventional open heart or minimally invasive techniques.

The KALIOS device is an adjustable annuloplasty ring, to be implanted by open surgery, having a hollow structure that comprises a flat rigid ring surrounding a deformable cage. The unique feature of KALIOS is that its annular shape and dimension can be finely adjusted percutaneously by an external actuator (three-balloon catheter) independently in the three areas corresponding to P1, P2 and P3

The primary objective of this clinical investigation is to assess the safety and effectiveness of KALIOS for the surgical treatment of Mitral Regurgitation with optional intra-operative and/or post-operative adjustment(s) The secondary objectives are to investigate the effects of KALIOS for the surgical treatment of Mitral Regurgitation on cardiac function and on patient functional status This clinical trial is prospective, non-randomized, single arm, multicentric & international. Up to 100 patients are expected to be enrolled to obtain 62 evaluable patients at one year,presenting with primary (degenerative) or secondary (functional) mitral valve regurgitation and who are candidate to a mitral valve repair.

ELIGIBILITY:
Inclusion Criteria:

- Patients must meet ALL the following inclusion criteria :

1. with primary or secondary mitral regurgitation recorded by TTE and confirmed during TEE where surgery for mitral valve repair is required with indications consistent with AHA/ACC and ESC/EACTS guidelines :

   1. primary (degenerative) : severe MR grade parameters (R Vol and EROA measured by PISA methods):

      * EROA regurgitant >60 ml and
      * Vena contracta width > 7mm and
      * Regurgitant fraction >50%
   2. Secondary (functional) : severe MR (EROA ≥30 mm²; R Vol > 30ml) may differ from the primary MR and are based on the prognostic value of these thresholds to predict the poor outcome, or for patients undergoing CABG
2. with LVEF ≥ 30%
3. in satisfactory condition, based on the physical examination and investigator's experience, with a life expectancy above one year after the intervention
4. with or without concomitant procedures as: CABG, other valve repair/replacement, pacemaker implantation, exclusion of left appendage (with device or surgically) and Maze (or PVI) procedure
5. willing to sign the informed consent;
6. able and willing to comply with all clinical investigation requirements, including the required study follow-up visits

Exclusion Criteria:

* Patients will be excluded if ANY of the following conditions are present:

  1. of age < 21 years;
  2. with echocardiographic measurements predicting SAM

     1. LVEDD < 45 mm
     2. C-Sd < 25mm (distance from the septum to the mitral valve coaptation point)
     3. Basal-IVDd > 15 mm
     4. aorto-mitral angle < 120°
     5. pre-repair posterior leaflet height > 15 mm
  3. with cardiogenic shock;
  4. with active endocarditis (or having had active endocarditis in the last three months);
  5. with active myocarditis;
  6. with heavily calcified mitral annulus;
  7. with mitral stenosis;
  8. unable to take anticoagulation medications;
  9. with a known untreatable allergy to contrast media or nickel;
  10. with a major or progressive non-cardiac disease that, in the investigator's experience, results in a life expectancy shorter than 1 year, or for whom the implant of the device produces an unacceptable increase of risk;
  11. with contraindication to transoesophageal echocardiography;
  12. with contraindication to cardiopulmonary bypass;
  13. who are pregnant or breast-feeding women;
  14. involved in any other clinical investigation for drugs or devices;
  15. unable to understand and sign the ICF in absence of legal protection;
  16. unable to read and write;

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of the effectiveness of KALIOS for the surgical treatment of Mitral Regurgitation with optional intra-operative and/or post-operative adjustment(s) | At 1 year
  Absence of Mitral Regurgitation of grade > 2 (through echographic assessment)
Assessment of the safety of KALIOS for the surgical treatment of Mitral Regurgitation with optional intra-operative and/or post-operative adjustment(s)Regurgitation with optional intra-operative and/or post-operative adjustment(s) | At 1 year
  Incidence of Major Adverse Cardiac Events (MACE)

SECONDARY OUTCOMES:
Assessment of the effectiveness of KALIOS for the surgical treatment of Mitral Regurgitation with optional intra-operative and/or post-operative adjustment(s) at each follow up | at 1, 3 6, 24, 36, 48 and 60 months
  Absence of Mitral Regurgitation of grade > 2 (through echographic assessment)
Assessment of the adjustment functionality of the device | immediately after annuloplasty, at 1, 3, 6, 12, 24, 36, 48 and 60 months
  Assessment of mitral leaflets coaptation (through echographic assessment)
Assessment of the adjustment functionality of the device | after any optional adjustment(s) performed immediately after annuloplasty, or following follow up visits at 1, 3, 6, 12, 24, 36, 48 and 60 months
  Assessment of the increase of mitral leaflets coaptation length (through echographic assessment)
Assessment of the safety of KALIOS for the surgical treatment of Mitral Regurgitation with optional intra-operative and/or post-operative adjustment(s)at each follow up | at 1, 3, 6, 24, 36, 48 and 60 months
  Incidence of Major Adverse Cardiac Events (MACE)

CONTACTS AND LOCATIONS:
Locations (9):
- Medical University of Vienna - Department of Surgery, Division of Cardiac Surgery, Vienna, Austria
- Germany (2):
  - University Clinic of Cardiac Surgery, Heart Center, Leipzig
  - Klinikum Passau, Passau
- Italy (5):
  - Maria Cecilia Hospital Cotignola, Cotignola
  - Careggi Hospital, Florence
  - Humanitas Research Hospital, Milan
  - Ospedale Luigi Sacco, Milan
  - Maria Eleonora Hospital Palermo, Palermo
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland